CLINICAL TRIAL: NCT03378713
Title: Clinical Effect of Follicular Preparation With Testosterone in Poor Ovarian Response: a Randomized Controlled Clinical Trial (TESTOPRIM)
Brief Title: Clinical Trial to Assess the Effect of Testosterone in Patients With Poor Ovarian Response (TESTOPRIM)
Acronym: TESTOPRIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TESTOPRIM
Record Dates: First submitted 2017-11-30; First posted 2017-12-20 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-02

CONDITIONS: Infertility, Female
Keywords: Poor Ovarian Response
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP 1: Long testosterone (Experimental): Application of testosterone in transdermal gel during the 2 cycles prior to initiation of controlled ovarian stimulation and until the onset of second menstruation (approximately 56 days). The COS begins the day after the last testosterone application.
  Interventions: Drug: GROUP 1: Long testosterone
- GROUP 2: Short testosterone (Active Comparator): Application of testosterone in transdermal gel begins on day 21 of menstrual cycle, from the luteal phase of the cycle prior to initiation of controlled ovarian stimulation and until menstruation (approximately 10 days). The COS begins the day after the last testosterone application.
  Interventions: Drug: GROUP 2: Short testosterone
- GROUP 3: Control (Active Comparator): The COS starts directly on the second day of the cycle without prior medication.
  Interventions: Drug: GROUP 3: Control

INTERVENTIONS:
Drug: GROUP 1: Long testosterone — Application of testosterone in transdermal gel during the 2 cycles prior to initiation of controlled ovarian stimulation and until the onset of second menstruation (approximately 56 days). The COS begins the day after the last testosterone application
  Arms: GROUP 1: Long testosterone
Drug: GROUP 2: Short testosterone — Application of testosterone in transdermal gel begins on day 21 of menstrual cycle, from the luteal phase of the cycle prior to initiation of controlled ovarian stimulation and until menstruation (approximately 10 days). The COS begins the day after the last testosterone application.
  Arms: GROUP 2: Short testosterone
Drug: GROUP 3: Control — The COS starts directly on the second day of the cycle without prior medication.
  Arms: GROUP 3: Control

SUMMARY:
Trial to determine the absolute and relative efficacy of two follicular preparation regimens with transdermal testosterone during the cycle (s) prior to the initiation of COS (controlled ovarian stimulation) in patients diagnosed with POR (poor ovarian response) for the increase in the number of mature oocytes recovered.

DETAILED DESCRIPTION:
POR is a challenge for reproductive medicine because of its impact on treatment outcomes and the lack of sufficiently proven therapeutic tools. According to recent publications based on retrospective studies of large registries, there is a correlation between the number of oocytes and LBR (live birth rate), so the investigators consider that variable mature oocytes are a reasonable compromise and a solid substitute for other outcome variables such as LBR or CPR (clinical pregnancy rate).

Regarding the duration of treatment, the investigators decided to include two groups of testosterone treatment (compared to the control group) with different duration. One will explore the role of testosterone in prolonged treatments (two full menstrual cycles). The other will test the pattern most commonly used in most studies, that is, testosterone in luteal phase of the previous cycle (about 10 days in short protocol with GnRH antagonist). In this way the investigators will establish an absolute comparison with the control group and relative between both treatment groups (long testosterone vs. short testosterone) to determine if / which of the two regimen (the two, only one or none) improves the number of mature oocytes recovered.

The product under investigation is testosterone gel, transdermal administration, 50 mg / single dose (Testim®, Ferring, Madrid, Spain). Regarding the dose, the investigators decided to keep the most used in the rest of studies (12.5 mg / day).

This study population will include only patients diagnosed with POR based on ESHRE Bologna criteria, in order to homogenize the population and allow comparisons with other studies in the future.

Regarding the dose, the investigators decided to keep the most used in the rest of studies (12.5 mg/day) which so far has been the only one proven effective. It is clearly possible that lower and more physiological doses are equally effective, but this yet has to be proven in well-designed studies. The gel is self-administered by the patients who are adequately instructed by a research nurse.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent prior to the completion of any procedure related to the clinical trial.
* Female older than 18 years old at the time of randomization.
* Prior diagnosis of poor ovarian response (POR) according to ESHRE Bologna criteria. Patients must meet at least 2 of the following:

  * Advanced maternal age (40 years or more) or any other risk factor for POR.
  * A previous POR (3 oocytes or less) with a conventional ovarian stimulation protocol.
  * Abnormal ovarian reserve test (RFA <5-7 or AMH 3.3-7.9 pmol / l).

Exclusion Criteria:

* Presence of uterine malformations, corrected or not.
* Presence of uterine pathology defined as submucous myomas or endometrial polyps, documented by transvaginal ultrasound.
* Couples with severe male factor defined as REM <1 or azoospermia.
* Hydrosalpinx unilateral or bilateral uncorrected.
* Perimenopausal patients with irregular menstrual cycles.
* Concurrent untreated endocrine disorders.
* Patients who have participated in a clinical trial in a period of less than one month.
* Known allergy to the drug.
* Patients who have received androgen treatment within 3 months prior to inclusion in the study.
* BMI> 35 kg / m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the trial treats female infertility
Enrollment: 63 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Total number of mature oocytes obtained at follicular puncture. | 36 hours after induction of ovulation with recombinant HCG.
  Determining whether a Follicular preparation with transdermal testosterone increases the number of mature oocytes retrieved in patients diagnosed with Poor Ovarian Response and which testosterone administration regimen is more effective for this purpose.

SECONDARY OUTCOMES:
Number of obtained embryos | 6 days after ovarian puncture.
Number of antral follicles at the start of stimulation | Time E: prior to controlled ovarian stimulation (at the beginning of the third cycle after inclusion and randomization, approximately 56 days after Day 0)
Initiation rate | Time E: prior to controlled ovarian stimulation (at the beginning of the third cycle after inclusion and randomization, approximately 56 days after Day 0)
  Quotient between the number of patients initiating COS and the total number of patients, overall and in each group
Number of days of stimulation duration | Time P (time of follicular puncture): 36 hours after the induction
Number of total follicles and greater than 16 mm | Time I (Day of induction): 10-12 days after controlled ovarian stimulation
Total dose of gonadotrophins used | Time I (Day of induction): 10-12 days after controlled ovarian stimulation
Cancellation rate due to lack of ovarian response | Time C: 10-12 days after controlled ovarian stimulation
Number of cumulus-oocyte complexes recovered on day of follicular puncture | Time P (time of follicular puncture): 36 hours after the induction
Fertilization rate | 24 hours after the puncture
Rate of cycles that achieve embryo transfer | Time ET ( day of embryo transfer): 4-5 days after the stimulation
Number of good quality embryos available | 48-72 hours after puncture
Number of embryos transferred | Time ET (day of embryo transfer): 4-5 days after the stimulation
Number of cycles with supernumerary embryos to freeze | 6 days after embryo transfer
Ongoing pregnancy rate per cycle started and per transfer | 70-75 days after embryo transfer
Clinical pregnancy rate per cycle started and per transfer | 30-35 days after embryo transfer
Miscarriage rate | At 11-13 weeks of pregnancy, if there is no previous news of the patient (Trial completion time)
Serum hormone levels | Day 0; Time I (day of induction): 10-12 days after controlled ovarian stimulation; and Time E (prior to controlled ovarian stimulation: at the beginning of the third cycle after inclusion and randomization, approximately 56 days after Day 0)
  Serum hormone levels of FSH, LH, E2, progesterone, testosterone, androstenedione, DHEA, SHBG and FAI

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Subirá, Principal Investigator — Hospital Universitari i Politècnic La Fe, Valencia, Spain
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tarlatzis BC, Zepiridis L, Grimbizis G, Bontis J. Clinical management of low ovarian response to stimulation for IVF: a systematic review. Hum Reprod Update. 2003 Jan-Feb;9(1):61-76. doi: 10.1093/humupd/dmg007. PMID 12638782
- [Background] Gorgy A, Naumann N, Bates S, Craft IL. Assisted conception following poor ovarian response to gonadotrophin stimulation. Br J Obstet Gynaecol. 1997 Dec;104(12):1420-1. doi: 10.1111/j.1471-0528.1997.tb11020.x. No abstract available. PMID 9422028
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Kyrou D, Kolibianakis EM, Venetis CA, Papanikolaou EG, Bontis J, Tarlatzis BC. How to improve the probability of pregnancy in poor responders undergoing in vitro fertilization: a systematic review and meta-analysis. Fertil Steril. 2009 Mar;91(3):749-66. doi: 10.1016/j.fertnstert.2007.12.077. Epub 2008 Jul 21. PMID 18639875
- [Background] Pandian Z, McTavish AR, Aucott L, Hamilton MP, Bhattacharya S. Interventions for 'poor responders' to controlled ovarian hyper stimulation (COH) in in-vitro fertilisation (IVF). Cochrane Database Syst Rev. 2010 Jan 20;(1):CD004379. doi: 10.1002/14651858.CD004379.pub3. PMID 20091563
- [Background] Jeve YB, Bhandari HM. Effective treatment protocol for poor ovarian response: A systematic review and meta-analysis. J Hum Reprod Sci. 2016 Apr-Jun;9(2):70-81. doi: 10.4103/0974-1208.183515. PMID 27382230
- [Background] Bastu E, Buyru F, Ozsurmeli M, Demiral I, Dogan M, Yeh J. A randomized, single-blind, prospective trial comparing three different gonadotropin doses with or without addition of letrozole during ovulation stimulation in patients with poor ovarian response. Eur J Obstet Gynecol Reprod Biol. 2016 Aug;203:30-4. doi: 10.1016/j.ejogrb.2016.05.027. Epub 2016 May 24. PMID 27236602
- [Background] Ertzeid G, Storeng R. The impact of ovarian stimulation on implantation and fetal development in mice. Hum Reprod. 2001 Feb;16(2):221-5. doi: 10.1093/humrep/16.2.221. PMID 11157810
- [Background] Van der Auwera I, D'Hooghe T. Superovulation of female mice delays embryonic and fetal development. Hum Reprod. 2001 Jun;16(6):1237-43. doi: 10.1093/humrep/16.6.1237. PMID 11387298
- [Background] Baker VL, Brown MB, Luke B, Smith GW, Ireland JJ. Gonadotropin dose is negatively correlated with live birth rate: analysis of more than 650,000 assisted reproductive technology cycles. Fertil Steril. 2015 Nov;104(5):1145-52.e1-5. doi: 10.1016/j.fertnstert.2015.07.1151. Epub 2015 Aug 18. PMID 26297646
- [Background] Escriva AM, Diaz-Garcia C, Monterde M, Rubio JM, Pellicer A. Antral Follicle Priming Before Intracytoplasmic Sperm Injection in Previously Diagnosed Low Responders: A Randomized Controlled Trial (FOLLPRIM). J Clin Endocrinol Metab. 2015 Jul;100(7):2597-605. doi: 10.1210/jc.2015-1194. Epub 2015 May 8. PMID 25955224
- [Background] Fanchin R, Cunha-Filho JS, Schonauer LM, Kadoch IJ, Cohen-Bacri P, Frydman R. Coordination of early antral follicles by luteal estradiol administration provides a basis for alternative controlled ovarian hyperstimulation regimens. Fertil Steril. 2003 Feb;79(2):316-21. doi: 10.1016/s0015-0282(02)04574-0. PMID 12568840
- [Background] Bosdou JK, Venetis CA, Kolibianakis EM, Toulis KA, Goulis DG, Zepiridis L, Tarlatzis BC. The use of androgens or androgen-modulating agents in poor responders undergoing in vitro fertilization: a systematic review and meta-analysis. Hum Reprod Update. 2012 Mar-Apr;18(2):127-45. doi: 10.1093/humupd/dmr051. Epub 2012 Feb 3. PMID 22307331
- [Background] Massin N, Cedrin-Durnerin I, Coussieu C, Galey-Fontaine J, Wolf JP, Hugues JN. Effects of transdermal testosterone application on the ovarian response to FSH in poor responders undergoing assisted reproduction technique--a prospective, randomized, double-blind study. Hum Reprod. 2006 May;21(5):1204-11. doi: 10.1093/humrep/dei481. Epub 2006 Feb 13. PMID 16476678
- [Background] Balasch J, Fabregues F, Penarrubia J, Carmona F, Casamitjana R, Creus M, Manau D, Casals G, Vanrell JA. Pretreatment with transdermal testosterone may improve ovarian response to gonadotrophins in poor-responder IVF patients with normal basal concentrations of FSH. Hum Reprod. 2006 Jul;21(7):1884-93. doi: 10.1093/humrep/del052. Epub 2006 Mar 3. PMID 16517559
- [Background] Fabregues F, Penarrubia J, Creus M, Manau D, Casals G, Carmona F, Balasch J. Transdermal testosterone may improve ovarian response to gonadotrophins in low-responder IVF patients: a randomized, clinical trial. Hum Reprod. 2009 Feb;24(2):349-59. doi: 10.1093/humrep/den428. Epub 2008 Dec 3. PMID 19054777
- [Background] Kim CH, Howles CM, Lee HA. The effect of transdermal testosterone gel pretreatment on controlled ovarian stimulation and IVF outcome in low responders. Fertil Steril. 2011 Feb;95(2):679-83. doi: 10.1016/j.fertnstert.2010.07.1077. PMID 20801436
- [Background] Kim CH, Ahn JW, Moon JW, Kim SH, Chae HD, Kang BM. Ovarian Features after 2 Weeks, 3 Weeks and 4 Weeks Transdermal Testosterone Gel Treatment and Their Associated Effect on IVF Outcomes in Poor Responders. Dev Reprod. 2014 Sep;18(3):145-52. doi: 10.12717/DR.2014.18.3.145. PMID 25949183
- [Background] Bosdou JK, Venetis CA, Dafopoulos K, Zepiridis L, Chatzimeletiou K, Anifandis G, Mitsoli A, Makedos A, Messinis IE, Tarlatzis BC, Kolibianakis EM. Transdermal testosterone pretreatment in poor responders undergoing ICSI: a randomized clinical trial. Hum Reprod. 2016 May;31(5):977-85. doi: 10.1093/humrep/dew028. Epub 2016 Mar 7. PMID 26956551
- [Background] Vendola KA, Zhou J, Adesanya OO, Weil SJ, Bondy CA. Androgens stimulate early stages of follicular growth in the primate ovary. J Clin Invest. 1998 Jun 15;101(12):2622-9. doi: 10.1172/JCI2081. PMID 9637695
- [Background] Weil S, Vendola K, Zhou J, Bondy CA. Androgen and follicle-stimulating hormone interactions in primate ovarian follicle development. J Clin Endocrinol Metab. 1999 Aug;84(8):2951-6. doi: 10.1210/jcem.84.8.5929. PMID 10443703
- [Background] Sen A, Hammes SR. Granulosa cell-specific androgen receptors are critical regulators of ovarian development and function. Mol Endocrinol. 2010 Jul;24(7):1393-403. doi: 10.1210/me.2010-0006. Epub 2010 May 25. PMID 20501640
- [Background] Nielsen ME, Rasmussen IA, Kristensen SG, Christensen ST, Mollgard K, Wreford Andersen E, Byskov AG, Yding Andersen C. In human granulosa cells from small antral follicles, androgen receptor mRNA and androgen levels in follicular fluid correlate with FSH receptor mRNA. Mol Hum Reprod. 2011 Jan;17(1):63-70. doi: 10.1093/molehr/gaq073. Epub 2010 Sep 14. PMID 20843821
- [Background] Walters KA. Role of androgens in normal and pathological ovarian function. Reproduction. 2015 Apr;149(4):R193-218. doi: 10.1530/REP-14-0517. Epub 2014 Dec 16. PMID 25516989
- [Background] Fooladi E, Reuter SE, Bell RJ, Robinson PJ, Davis SR. Pharmacokinetics of a transdermal testosterone cream in healthy postmenopausal women. Menopause. 2015 Jan;22(1):44-9. doi: 10.1097/GME.0000000000000259. PMID 24845394
- [Background] Sunkara SK, Rittenberg V, Raine-Fenning N, Bhattacharya S, Zamora J, Coomarasamy A. Association between the number of eggs and live birth in IVF treatment: an analysis of 400 135 treatment cycles. Hum Reprod. 2011 Jul;26(7):1768-74. doi: 10.1093/humrep/der106. Epub 2011 May 10. PMID 21558332
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Fertility: Assessment and Treatment for People with Fertility Problems. London: Royal College of Obstetricians & Gynaecologists; 2013 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK247932/ PMID 25340218